CLINICAL TRIAL: NCT05838521
Title: A Phase II Evaluation of Sacituzumab Govitecan (IMMU-132), an Anti-Trop-2-SN-38 Antibody-drug Conjugate in Patients With Recurrent or Persistent Cervical Cancer
Brief Title: A Study of Sacituzumab Govitecan (IMMU-132) in Patients With Recurrent or Persistent Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000023639
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Govitecan (Experimental): Sacituzumab govitecan, 10 mg/kg for the first 2 weeks of 21-day cycle until progression or adverse effects prohibit further treatment.
  Interventions: Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Sacituzumab govitecan — This is a non-randomized Phase 2 study of sacituzumab govitecan (IMMU-132).
  Other Names: Trodelvy

SUMMARY:
This is a non-randomized Phase 2 study of sacituzumab govitecan (IMMU-132) in subjects with recurrent or persistent cervical cancer.

DETAILED DESCRIPTION:
This is an open-label, Phase 2 study designed to assess the clinical activity of sacituzumab govitecan in subjects with recurrent or persistent cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiologically confirmed (i.e., CAT scan and/or MRI) persistent or recurrent histologically confirmed cervical cancer of epithelial origin who have progressed following at least one prior chemotherapy treatment regimen.

  * Must have availability of archival tumor tissue FFPE block for TROP-2 testing
  * Chemotherapy administered concurrent with primary radiation (i.e., weekly cisplatin) is not counted as a systemic chemotherapeutic regimen for management of persistent or recurrent carcinoma of the cervix.
* All patients must have measurable disease.
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST v1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence following completion of radiation therapy.
* Patients with measurable recurrent disease of any previous substage (I-IV) are eligible to enrollment.
* Patients must have adequate bone marrow function: WBC greater than or equal to 3,000/ul, Platelets greater than or equal to 75,000/ul, Granulocytes greater than or equal to 1500/ul.
* Patients must have adequate renal function: creatinine less than or equal to 2.0 mg/dL.
* Patients must have adequate hepatic function: bilirubin ≤ 1.5 institutional upper limit of normal, aspartate aminotransferase [AST], and alanine aminotransferase [ALT] ≤ 2.5 × IULN or ≤ 5 × IULN if known liver metastases
* Patients must have an ECOG performance status of 0 or 1.
* Patients must have signed an approved informed consent.
* Patients must be at least 2 weeks beyond prior treatment (chemotherapy, investigational drugs including small molecular inhibitors, endocrine therapy, immunotherapy and/or radiation therapy) or major surgery.
* Patients must be at least 2 weeks beyond high dose systemic corticosteroids (however, low dose corticosteroids < or equal to 20 mg prednisone or equivalent daily are permitted)
* Patients must have recovered from all acute toxicities to Grade 1 or less from adverse events due to a previously administered agent Note: Patients with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients with recurrent disease may have received no more than 2 prior chemotherapies for treatment of their cervical cancer.
* Patients may have received prior immunotherapy therapy alone or in combination with chemotherapy. A 4-week washout period is required between prior immunotherapy treatment and first dose of sacituzumab govitecan.
* Patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the study entry and be practicing an effective form of contraception during the study and until conclusion of 12-week post-treatment evaluation period.
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Patients with a positive serum pregnancy test or women who are breastfeeding.
* Patients with known hypersensitivity to the study drug, its metabolites, or formulation excipient.
* Patients who require ongoing therapy with or prior use of any prohibited medication(s) such as UGT1A1 inhibitors.
* Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
* Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the patient's participation in the study.
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancers or carcinoma in situ of the cervix, are excluded if there is any evidence of other malignancy being present within the last 5 years.
* Patients with a significant history of cardiac disease within 6 months, i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure (NYHA classification III-IV) or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring antiarrhythmia therapy.
* Patients with known history of clinically significant active COPD, or other moderate-to-severe chronic respiratory illness present within 6 months
* Patients with any unstable medical issue (including cardiac issues as above, active treatment for symptomatic pulmonary embolism, CVA, renal or hepatic insufficiency, and active infection/sepsis requiring IV antibiotics).
* Have known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to the first dose of study drug and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are taking ≤20 mg/day of prednisone or its equivalent. All patients with carcinomatous meningitis are excluded regardless of clinical stability
* Patients who have an uncontrolled seizure disorder, or active neurological disease.
* Have known history of HIV-1 or 2 (or positive HIV-1/2 antibody) with detectable viral load OR taking medications that may interfere with SN-38 metabolism
* Have active HBV or HCV. In subjects with a history of HBV or HCV, subjects with a detectable viral load will be excluded.
* Known hemorrhagic diathesis or active bleeding disorder.
* Patients with Gilbert's disease
* Presence of bulky disease (defined as any single mass >7 cm in its greatest dimension). Patients with a mass over 7 cm, but otherwise eligible, may be considered for enrollment after discussion and approval with the study PI.
* Patients with active ≥ grade 2 anorexia, nausea or vomiting, and/or signs of intestinal obstruction.
* Prior history of intestinal obstruction within 6 months of initiation of study treatment.
* Patients with a history of an anaphylactic reaction to irinotecan or ≥ Grade 3 toxicity to prior irinotecan.
* Have previously received topoisomerase I inhibitors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 4 Years
  Objective response rate (complete response and partial response rates) by RECIST1.1 criteria in patients with recurrent or persistent cervical cancer.

SECONDARY OUTCOMES:
Duration of overall survival (OS) | 6 Years
  Overall survival is defined as the duration of time from study entry to death or the date of last contact.
Duration of progression free survival (PFS) | 6 Years
  Progression free survival is defined as the duration of time from study entry to time of progression, death, or is censored at date of last disease assessment.
Durable disease control rate (DDCR) | 6 Years
  The percentage of patients who have achieved complete response, partial response, and stable disease.
Assess the safety profile of sacituzumab govitecan in cervical cancer patients (adverse events as assessed by CTCAE v5.0) | 6 Years
  Incidence of treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D. Santin, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Cleveland Clinic, Cleveland, Ohio